CLINICAL TRIAL: NCT05353465
Title: Cervicale Facet Joint Denervation With a Trident Electrode, a Retrospective Observational Study
Brief Title: The Cervical Trident Study
Status: Completed | Type: Observational
Sponsor: Ospedale Regionale di Lugano (Other)
Responsible Party: Principal Investigator, Eva Koetsier MD PhD LLM, Pain Management Center, Neurocenter of Southern Switzerland, EOC, Ospedale Regionale di Lugano
Other Study IDs: The Cervical Trident Study
Record Dates: First submitted 2022-04-23; First posted 2022-04-29 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Facet Joint Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Radiofrequency denervation of the cervical facet joint — Radiofrequency denervation of the medial branch of the dorsal ramus of the cervical facet joint with a three-tined expandable needle.

SUMMARY:
This observational retrospective study evaluates the efficacy of RF with the three-tined expandable electrode needle compared to before treatment in the treatment of chronic cervical facet joint pain.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Patients with neck pain
* Patient who had two diagnostic medial branch blocks with significant (>50%) improvement on both injections.

Exclusion Criteria:

- No patient related outcome measures available in hospital's patient charts

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All adult patients that are treated with radiofrequency (RF) ablation of the facet joints in patients selected by symptom improvement with dual medial branch blocks.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2022-05-20 (Actual); Primary Completion 2022-06-03 (Actual); Study Completion 2022-07-03 (Actual)

PRIMARY OUTCOMES:
Pain measurement by numeric rating score | 2 months after injection in comparison to baseline
  The primary outcome of this study is pain measured with the numeric rating score (NRS): 11-point NRS ranging from 0 (no pain at all) to 10 (the worst imaginable pain). A score of zero (0) will indicate that the patient is pain free, while a score of ten (10) will indicate that they are experiencing the worst pain imaginable.

SECONDARY OUTCOMES:
Patient Global Impression of Change (PGIC) | 2 months after injection
  The PGIC rating is increasingly being used for determining clinically important change in measures such as ratings of pain. This scale is designed to quantify patient's improvement or deterioration over time, usually either to determine the effect of an intervention or to chart the clinical course of a condition. The scales ask that a person assess his or her current pain, recall that status at a previous time-point, and then calculate the difference between the two.
  * very much improved
  * much improved
  * minimally improved
  * no change
  * minimally worse
  * much worse
  * very much worse
Use of analgesics | 2 months after injection
  The quantity of analgesics that the patient assumes for the pain:
  * All stopped
  * Decreased
  * Equal
  * Increased
Sleep | 2 months after injection
  Question: 'your sleep quality is:
  * Improved
  * Equal
  * Worsened'
Walking ability | 2 months after injection
  Question: 'after the treatment, you can walk:
  * More than before
  * Same as before
  * Less than before'
Patient satisfaction | 2 months after injection
  Question: are you satisfied with the result: YES/NO

CONTACTS AND LOCATIONS:
Overall Officials: Eva Koetsier, MD PhD LLM, Principal Investigator — Neurocenter of Southern Switzerland, EOC, Lugano
Locations (1):
- Pain Management Center, Neurocenter of Southern Switzerland, Lugano, Switzerland

IPD SHARING:
Plan to Share IPD: No